CLINICAL TRIAL: NCT05682755
Title: Chidamide Prevents the Recurrence of High-risk Acute Myeloid Leukemia After Allogeneic Hematopoietic Stem-cell Transplantation: A Prospective, Single-centered, Single-arm, Phase I/II Clinical Study
Brief Title: Chidamide Prevents Recurrence of High-risk AML After Allo-HSCT
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sichuan University (Other)
Responsible Party: Principal Investigator, Jie Ji, Principle Investigator, Sichuan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTChi 1.0
Record Dates: First submitted 2022-12-27; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2022-12

CONDITIONS: Leukemia, Myeloid, Acute
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Chidamide (Experimental)
  Interventions: Drug: Chidamide

INTERVENTIONS:
Drug: Chidamide — initial time：platelet count ≥50×10^9/L after allo-HSCT initial dose: 5 mg oral twice weekly initial adjustment: according to the platelet count tested weekly platelet count ≥50×10^9/L-increased by 5 mg 20×10^9/L≤ platelet count <50×10^9/L-remains unchanged platelet count <50×10^9/L- reduced by 5 mg maximum dose: 20 mg oral twice weekly terminal time: 180 days after allo-HSCT

SUMMARY:
The goal of this phase I/II clinical trial is to test in high-risk acute myeloid leukemia (AML) patients undergoing allogeneic hemopoietic stem-cell transplantation (allo-HSCT). The main question it aims to answer is:

• The efficacy and safety of chidamide maintenance therapy in reducing the recurrence rate and GVHD incidence in high-risk AML patients after allo-HSCT.

Participants will take oral chidamide (Epidaza) until 180 days after allo-HSCT.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old and ≤ 65 years old when signing the Informed Consent Form (ICF);
2. KPS score > 60 or ECOG score 0-2;
3. The expected survival period > 3 months;
4. Received allo-HSCT and achieved complete remission (CR);
5. Reach the standard of hematopoietic reconstitution (neutrophil count ≥ 0.5×10^9/L for 3 consecutive days without G-CSF application, platelet count ≥ 20×10^9/L for 7 consecutive days without platelet transfusion, Hb ≥ 80 g /L without red blood cell transfusion); and neutrophil count ≥ 1.5×10^9/L, platelet count ≥ 50×10^9/L within 45 days after transplantation;
6. No central nervous system involvement or clinical symptoms after transplantation;
7. Those who have no serious functional damage to important organs of the body;
8. Fully understand and be informed of this study and sign the ICF; willing to follow and have the ability to complete all test procedures;
9. Females of childbearing age must afford a serum pregnancy test within 7 days before the first dose, and the result should be negative; female participants and their partners should agree to use effective contraception from signing the ICF until 6 months after the last dose.

Exclusion Criteria:

1. Serious basic diseases of important organs: such as myocardial infarction, chronic cardiac insufficiency, decompensated hepatic insufficiency, renal function, gastrointestinal insufficiency, etc.;
2. Uncontrolled active infection (including bacterial, fungal, or viral infection), and drug treatment is ineffective;
3. Participating in other clinical studies, or planning to start treatment in this study and less than 4 weeks before the end of treatment in the previous clinical study;
4. Poor graft function (PGF) occurred after allo-HSCT;
5. Combined with other malignant tumors and require treatment;
6. Active GVHD;
7. Have a history of allergy to Chidamide;
8. Pregnant or lactating females;
9. Patients with known history of human immunodeficiency virus (HIV) virus infection and/or acquired immunodeficiency syndrome;
10. Patients with active chronic hepatitis B or active hepatitis C;
11. History of prolonged QT syndrome;
12. Patients considered by other researchers to be unsuitable for this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Estimated)
Dates: Start 2022-12-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 2 years
  Progression free survival of this group of patients at the end of 2 year

SECONDARY OUTCOMES:
100 day adverse events (AE) | Day +100
  non-hematologic adverse events
Non-relapse mortality (NRM) | 6 months
  Non-relapse mortality of this group of patients at the end of 6 month
Overall survival (OS) | 2 years
  Overall survival of this group of patients at the end of 2 year
Relapse rate | 2 years
  Relapse rate of this group of patients at the end of 2 year
Cumulative incidence of acute graft versus host disease (aGVHD) | Day +100
  Cumulative incidence of acute graft versus host disease (aGVHD) of this group of patients at day+100
Cumulative incidence of chronic graft versus host disease (cGVHD) | 2 years
  Cumulative incidence of chronic graft versus host disease (cGVHD) of this group of patients at the end of 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital of Sichuan University, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes
Release after the publication of results of this trial
Supporting Information: Study Protocol
Time Frame: after the publication of results of this trial